CLINICAL TRIAL: NCT03695952
Title: A Prospective Cohort Study of Patients with Hepatobiliary Cancer Treated with Immune Checkpoint Inhibitors
Status: Active, not recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Assistant Professor, Asan Medical Center
Other Study IDs: ICI_Biomarker
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma; Biliary Tract Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms | interventions — Nivolumab; pembrolizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hepatocellular carcinoma: Hepatocellular carcinoma patients treated with nivolumab
  Interventions: Drug: Nivolumab or pembrolizumab
- Biliary Tract Cancer: Biliary tract cancer patients treated with pembrolizumab
  Interventions: Drug: Nivolumab or pembrolizumab

INTERVENTIONS:
Drug: Nivolumab or pembrolizumab — Nivolumab 3 mg/kg intravenous every 2 weeks; Pembrolizumab 200 mg intravenous every 3 weeks
  Other Names: Immune checkpoint inhibitors

SUMMARY:
Although immune checkpoint inhibitors including nivolumab and pembrolizumab are now available for the management of hepatobiliary cancers in Korea, there is a lack of data for the efficacy and safety of these agents in the real-world setting. This study aims to prospectively evaluate the efficacy of safety of nivolumab and pembrolizumab against advanced hepatocellular carcinoma and biliary tract cancer.

DETAILED DESCRIPTION:
Nivolumab 3 mg/kg intravenous every 2 weeks has been recently approved by US FDA for the management of patients with sorafenib-failed advanced HCC based on the promising data of Checkmate-040 phase I/II study. Although there is a lack of prospective data for pembrolizumab in biliary tract cancer except for small phase 1 trial, pembrolizumab is now available for use in Korea for the management of advanced biliary tract cancer. Because the approval of these agents was based on the small sample size, further prospective evaluation of nivolumab or pembrolizumab in patients with hepatobiliary cancer is needed.

ELIGIBILITY:
Inclusion Criteria:

* Biliary tract cancer (intrahepatic or extrahepatic cholangiocarcinoma and gallbladder cancer) or hepatocellular carcinoma
* Planned immune checkpoint inhibitors including nivolumab or pembrolizumab
* Written informed consent

Exclusion Criteria:

* Not available for the treatment with immune checkpoint inhibitors

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatobiliary cancer patients treated with nivolumab or pembrolizumab
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 months
  Proportion of complete response and partial response according to the Response Evaluation Criteria in Solid Tumors version 1.1

SECONDARY OUTCOMES:
Adverse events | 6 months
  Toxicity of nivolumab or pembrolizumab according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Changhoon Yoo, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuah S, Lee J, Song Y, Kim HD, Wasser M, Kaya NA, Bang K, Lee YJ, Jeon SH, Suthen S, A'Azman S, Gien G, Lim CJ, Chua C, Hazirah SN, Lee HK, Lim JQ, Lim TKH, Yeong J, Chen J, Shin EC, Albani S, Zhai W, Yoo C, Liu H, Choo SP, Tai D, Chew V. Uncoupling immune trajectories of response and adverse events from anti-PD-1 immunotherapy in hepatocellular carcinoma. J Hepatol. 2022 Sep;77(3):683-694. doi: 10.1016/j.jhep.2022.03.039. Epub 2022 Apr 15. PMID 35430299